CLINICAL TRIAL: NCT05465018
Title: Performance Assessment Study VitalSigns Camera
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Philips Clinical & Medical Affairs Global (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ICBE-S-000822
Record Dates: First submitted 2022-07-15; First posted 2022-07-19 (Actual); Last update posted 2022-08-18 (Actual); Status verified 2022-08

CONDITIONS: Healthy Humans; Vital Signs Monitoring
Keywords: Pulse rate; Remote Photoplethysmography; Algorithms
MeSH Terms: interventions — Masks

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Healthy volunteers (Experimental): 1 arm. Healthy volunteers assigned to different interventions
  Interventions: Device: Happy Flow / Baseline; Device: Make-up; Device: Sunglasses; Device: Face mask; Device: Minimum requirements camera; Device: Worst case hardware; Device: Damaged lens; Device: Face or chest outside test frame

INTERVENTIONS:
Device: Happy Flow / Baseline — Baseline (without make-up or mask)
Device: Make-up — To test device on participant who is wearing facial make-up
Device: Sunglasses — To test device on participant who is wearing sunglasses
Device: Face mask — To test device on participant who is wearing a facial mask
Device: Minimum requirements camera — To test the minimum requirements of the camera
Device: Worst case hardware — To test if software still works with an older smartphone
Device: Damaged lens — To test if software is still working when the lens of the smartphone is damaged
Device: Face or chest outside test frame — To test software if the participants face or chest is outside the test frame

SUMMARY:
This Performance Assessment Study will focus on testing the performance of the VitalSigns Camera under various suboptimal use cases. The software makes it possible to measure the pulse rate (PR) and respiration rate (RR) without the device being in contact with the subject. The software delivers fast and accurate results (in less than one minute). Vital signs camera (VSC) product will be used via a demonstrator app on one of the smartphones during the study sessions (camera of the phone will be used by the VSC product). Devices will be provided by the researchers.

The subject will be asked to perform a number of assignments with the software application. The study involves taking a number of measurements of the subject's PR using the VitalSigns Camera software application (which is installed on a smartphone or laptop). In this study only PR is measured and not RR as the latter parameter is not affected by the designed test cases. The total duration of the session will be approximately 1 hour. In total, approximately 30 healthy volunteers will participate in this study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteer must 18 years or older
* Participants willing to give informed consent
* Willingness to have vital signs measured by a medical mobile application
* Willingness to put on sunglasses
* Willingness to put on facial makeup
* Willingness to put on a face mask covering mouth and nose
* Willingness to sit still up to 2 minutes per measurement

Exclusion Criteria:

* Individuals who are not able to read and understand the English language
* Known allergic reaction to facial make-up
* COVID-19 exclusion criteria:

  * Currently displaying COVID-19-related symptoms, namely a fever, cough and/or difficulty breathing
  * Having been positively tested as infected with COVID-19 in the past 14 days
  * Travelled to or from high risk COVID-19 areas in the past 14 days
  * Been in contact with a (suspected) COVID-infected person in the past 14 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-07-07 (Actual); Primary Completion 2022-07-22 (Actual); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Primary endpoint | Each participants will have measurement for 1 hour on 1 day. Study will be completed within 1 week.
  To compare the Pulse Rate (Beats per Minute) measured by the VitalSigns Camera with the Pulse Rate measured by the reference device.

CONTACTS AND LOCATIONS:
Locations (1):
- Philips Research North America, Cambridge, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No